CLINICAL TRIAL: NCT01384604
Title: Neurophysiological and Genetic Studies in Schizophrenia and Other Psychiatric Disorders
Brief Title: Neurophysiological Studies in Schizophrenia and Psychiatric Disorders
Acronym: BSNIP
Status: Completed | Type: Observational
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Carol A. Tamminga, Principal Investigator, University of Texas Southwestern Medical Center
Other Study IDs: STU 112010-097; 1R01MH077851-01A2 (NIH)
Record Dates: First submitted 2011-06-27; First posted 2011-06-29 (Estimated); Last update posted 2019-01-16 (Actual); Status verified 2019-01

CONDITIONS: Schizophrenia; Schizoaffective Disorder; Bipolar Disorder
Keywords: Schizophrenia; Schizoaffective disorder; Bipolar disorder; Psychosis; Genetics; Phenotype
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Bipolar Disorder

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood, no more than 30cc; urine, small collection cup (about 30cc) to administer drug urine screen and pregnancy tests for females; buccal swabs (at least 5 swabs from volunteers that cannot donate blood); and, optional: 4mm punch of skin for dermal biopsy.
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The overall goal of this project is to identify intermediate phenotypes for psychosis across the schizophrenia and bipolar disorders boundary with implications for future genetic studies. Recent studies provide considerable evidence that schizophrenia and psychotic bipolar disorder may share overlapping etiologic determinants. Identifying disease-related genetic effects is a major focus in schizophrenia and bipolar research, with enormous implications for diagnosis and treatment for these two disorders. Efforts have been multifaceted, with the ultimate goal of describing causal paths from specific genetic variants, to changes in neuronal functioning, to altered brain anatomy, to behavioral and functional impairments. Parallel efforts have identified and refined several alternative endophenotypes that are stable, heritable, have (partly) known biological substrates, and are associated with psychosis liability. Although many such endophenotypes have been individually studied in schizophrenia, and to a lesser extent in bipolar disorder, no study has comprehensively assessed a broad panel of these markers in the two disorders with parallel recruitment, and the extent to which they mark independent aspects of psychosis risk, or their overlap in the two disorders. In this research project, we will examine a broad panel of putative endophenotypes in affected individuals and their first degree, biological relatives in order to: 1) characterize the degree of familial phenotypic overlap between schizophrenia and psychotic bipolar disorders; 2) identify patterns of endophenotypes unique to the two disorders; and, 3) contrast the heritability of endophenotypes across the disorders. We will obtain measures of neurophysiology (e.g., eye tracking, P50 gating, PPI, and P300), neurocognition (e.g., attention/vigilance, episodic and working memory), and brain structure (e.g., volumes of gray and white matter in specified brain regions). Blood samples will also be collected and stored for formal DNA linkage analyses using the independent phenotypes identified above. All volunteers will also be given the option to donate dermal biopsies for future research studies.

Establishing similarities and differences in the endophenotypic signatures within schizophrenia and bipolar families will provide important insights for future genetic studies, and clarify concepts about common and distinct aspects of pathophysiology, potentially meaningful heterogeneity with disorders, and the clinical boundaries of the two most common psychotic disorders in adult psychiatry. This line of investigation will potentially impact our conceptualization of psychotic disorders, help us make critical strides to identify the pathophysiology of psychosis, and guide development of new specific treatments targeting particular deficits.

ELIGIBILITY:
Inclusion Criteria:

* DSM-IV diagnosis of schizophrenia, schizoaffective disorder, or bipolar disorder with psychotic features
* Ages 15-70 years old
* Must have a first degree, biological relative in the same age range who is willing and available to participate

Exclusion Criteria:

* Diagnosis of an organic brain disease
* Meets criteria for alcohol or substance abuse with the last month; alcohol or substance dependence within the last 3 months; or, has an extensive history of drug dependence
* History of seizures, serious head injury, concussions, or other evidence of brain disease
* Medical illnesses that are not currently well-controlled

Ages: 15 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Individuals with schizophrenia, schizoaffective, or bipolar I disorder.
Sampling Method: Non-Probability Sample
Enrollment: 1189 (Estimated)
Dates: Start 2007-12; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Texas Southwestern Medical Center, Dallas, Texas, United States

REFERENCES:
- See also: UT Southwestern's "Find a Clinical Trial" Search (FaCT) — http://www.utsouthwestern.edu/utsw/cda/dept226287/files/308724.html